CLINICAL TRIAL: NCT03104283
Title: A Multicenter, Single-arm, Phase Ⅱ Clinical Trial of Apatinib Monotherapy in Elderly Patients With Advanced Gastric Cancer(GC)
Brief Title: Apatinib for the Elderly Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Professor, Affiliated Hospital of Qinghai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHQU-2017001
Record Dates: First submitted 2017-04-01; First posted 2017-04-07 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
Keywords: apatinib; gastric cancer; elderly patients
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Group (Experimental): take apatinib orally (500mg/d or 250mg/d, once a day, continuously )
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — take apatinib orally until disease progression or appearance of unbearable toxicity
  Other Names: Apatinib group

SUMMARY:
The purpose of our study is to assess the efficacy and safety of apatinib in elderly advanced gastric cancer patients, and to find the relationship between the expression of VEGFR-2 and efficacy of apatinib treatment.

DETAILED DESCRIPTION:
The trial is funded by Chinese Society of Clinical Oncology-Beijing Xisike Clinical Oncology Research Fundation. The trial is prepared to be registered on the clinicaltrail.gov.

Quality assurance plan: Every participant is enrolled or excluded by two practiced investigators. And two investigators participate in all steps of the trail, including the record of the data, which is compared by the investigators. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the staff of research and financial department of Affliated Hospital of Qinghai University.

Data check: The investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification: The investigators assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms.

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 47 participants to take part in the trail. The investigators can recruit about 20 participants every year according to previous experiences, so the investigators should recruit about two years.

Plan for missing data: The investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Statistical analysis plan: Statistical analyses would be performed by using SPSS software, version 13.0 (SPSS Inc., IL, USA). Survival analysis would be performed using Kaplan-Meier methodology. Fisher's exact test would be used to analyze the efficacy of treatment. Cox proportional hazards model would be used for multivariate analysis. The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients (aged ≥ 60 years) with histologically confirmed advanced adenocarcinoma of the stomach or gastroesophageal junction;
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
3. Progression with or intolerance to one or more lines of chemotherapy;
4. At least one measurable lesion as defined by RECIST 1.1;
5. With acceptable hematologic, cardiac, hepatic, pulmonary and renal function;
6. Can take apatinib orally;
7. Estimated life expectancy ≥ 3 months.

Exclusion Criteria:

1. Patients cannot take apatinib orally for any reason;
2. Patients with uncontrolled central nervous system (CNS) metastases;
3. Patients with massive hydrothorax or ascites;
4. Proteinuria 2+ or 24-hour urinary protein ≥ 1g;
5. Newly-happened traumatism or pathological fracture;
6. Estimated life expectancy ˂ 3 months;
7. Received chemotherapy in the past 28 days before enrollment;
8. Patients with uncontrolled blood pressure on medication (≥ 140/90 mmHg);
9. Patients with bleeding tendency, receiving thrombolytics or anticoagulants, receiving intravenous antibiotic treatment, had received bevacizumab or other VEGF TKIs before, or with other primary malignancy (except basal cell skin cancer or cervical carcinoma in situ).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  PFS was defined to be the time from registration to the date of disease progress sion or death resulting from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR was defined as the proportion of eligible patients who achieved a confirmed complete response(CR )or partial response (PR) by RECIST 1.1 criteria evaluated by the investigators.
Disease control rate (DCR) | 1 year
  DCR was defined as the proportion of patients who achieved CR, PR and stable disease (SD) for at least 8 weeks.
Overall survival (OS) | 1 year
  OS was defined to be the time from registration to the date of death resulting from any cause or the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jiuda Zhao, M.D., Principal Investigator — Affiliated Hospital of Qinghai University
Locations (5):
- China (5):
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - People's Hospital of Qinghai Province, Xining, Qinghai
  - Qinghai Red Cross Hospital, Xining, Qinghai
  - the Fifth People's Hospital of Qinghai Province, Xining, Qinghai
  - Yangquan No.1 People's Hospital, Yangquan, Shanxi